CLINICAL TRIAL: NCT02981355
Title: Randomized Evaluation of BST-CarGel Versus Microfracture Alone On Recovery From Distal Femoral Cartilage Lesions
Acronym: RECORD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Piramal Healthcare Canada Ltd (Industry)
Collaborators: Smith & Nephew, Inc. (Industry); Global Research Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BST-CarGel Pr001
Record Dates: First submitted 2016-11-21; First posted 2016-12-05 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2017-08

CONDITIONS: Traumatic; Lesion; Degenerative Lesion of Articular Cartilage of Knee
Keywords: BST-CarGel; Microfracture; Cartilage Lesion, Chondral Lesion; Femoral condyle; Bone Marrow Stimulation; Cartilage Repair; Tear of Articular Cartilage of Knee, Current
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microfracture treatment (Active Comparator): Microfracture surgery of the femoral condyle
  Interventions: Procedure: Microfracture treatment
- BST-CarGel plus microfracture treatment (Experimental): BST-CarGel combined with fresh, autologous whole blood and applied to the lesion on the femoral condyle with a syringe following an arthroscopic microfracture surgery.
  Interventions: Procedure: Microfracture treatment; Device: BST-CarGel

INTERVENTIONS:
Procedure: Microfracture treatment — Microfracture is performed by penetrating the subchondral bone beneath the cartilage lesion inducing a bleeding response.
Device: BST-CarGel — BST-CarGel is combined with fresh, autologous whole blood and applied to the lesion on the femoral condyle with a syringe following microfracture arthroscopic surgery.
  Arms: BST-CarGel plus microfracture treatment

SUMMARY:
This multi-centre randomized, controlled trial will assess the impact of BST-CarGel scaffold with microfracture versus microfracture alone on short and long term clinical benefit in patients with cartilage lesions of the femoral condyle requiring operative management.

DETAILED DESCRIPTION:
The current standard of treatment for cartilage lesions on the femoral condyle is microfracture, which is conducted by penetrating the subchondral bone below the lesion. This procedure creates a natural healing response as a result of the bleeding and clotting caused by the microfracture, restoring the lesion. BST-CarGel (Piramal Life Sciences, Bio-Orthopaedic Division), a liquid chitosan-containing polymer scaffolding, has been developed as an intra-articular injectable scaffold to aid in the stabilization of the blood clot created by microfracture. BST-CarGel does not interfere with the normal clotting process; however, it enables a prolonged healing time due to the increased stabilization of the clot within the lesion and the inhibition of clot retraction.

The RECORD trial is a multi-centre, randomized, controlled trial to assess the impact of the BST-CarGel scaffold and microfracture versus microfracture alone on short term clinical benefit as measured by loaded knee pain (single leg squat) on a visual analogue scale (3-6 months), mid-long term clinical benefit as measured by the same loaded knee pain (single leg squat) (9, 12, and 24 months) and Tegner Activity Score (TAS), International Knee Documentation Committee (IKDC), and Knee Injury and Osteoarthritis (KOOS) at 3, 6, 9, 12 and 24 months post-operatively. Approximately 158 participants with full-thickness grade III and IV cartilage lesions will be randomised in a 1:1 ratio to receive one of the two treatments during an arthroscopic procedure and will be followed for up to 24 months to collect outcomes.

ELIGIBILITY:
Inclusion Criteria:

* requires cartilage repair treatment due to distal femoral cartilage lesion
* is 18-55 years of age at the time of surgery
* has single, focal cartilage lesion on one of the femoral condyles
* has symptomatic cartilage lesion that has failed conservative management
* has a single lesion classified as focal, full-thickness grade 3 or 4 according to the ICRS (3A, 3B, 3C, 3D and 4A)
* an area of lesion between 1.5-3 cm2 after debridement
* has a stable knee (<5-mm side-to-side difference on Lachman and varus and valgus stress testing and grade 0 or 1 on the pivot-shift test) and an intact meniscal rim
* is willing and able to participate in required follow-up visits at the investigational site and to complete study procedures and questionnaires and recommended physiotherapy regimen
* has agreed to discontinue the use of all knee pain medication 3 days before the pre-treatment visit and the post-treatment follow-up visits at 3, 6, 9, 12, and 24 months
* has consented to participating in the study by signing the IRB/EC approved informed consent form
* no deep osteochondral defect ( < 5 mm bone loss)

Exclusion Criteria:

* has multiple lesions or kissing (opposing) lesion(s) greater than GII
* has clinically relevant compartment malalignment (>5°)
* has bone cyst(s) associated with, or adjacent to, the index lesion
* has Osteochondritis Dissecans with bone or bone-cartilage fragment in place
* has had ligament treatments in the index knee within the previous 24 months
* has had surgical cartilage treatments in the index knee within previous 12 months
* has had intra-articular injections in the index knee within the previous 2 months
* has diagnosis of an immunosuppressive disorder
* has a BMI > 30 kg/m2
* has concomitant healing bone fractures
* has a single lesion classified as focal, full-thickness grade 4B as defined by ICRS
* has noteworthy pain in the ipsilateral hip or ankle or contralateral hip, knee, or ankle
* has inflammatory arthropathy
* has blood clotting disorders, was receiving anticoagulant therapy, or has recurring deep vein thrombosis
* has a serious heart condition or liver and/or renal abnormalities diagnosed within the previous 24 months
* has chronic infection of the lower joint extremities
* has a history of alcohol or drug abuse within the previous 12 months
* is facing current or impending incarceration
* has a known allergy to shellfish
* is pregnant or plans to become pregnant during the course of the study
* in the opinion of the PI, has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, drug or alcohol abuse
* chronic knee pain
* has a documented medical history of vitamin-D deficiency that is not being managed with supplementation
* is entered in another investigational drug, biologic, or device study or has been treated with an investigational product in the past 30 days
* requires an open procedure
* is known to be at risk for lost to follow-up, or failure to return for scheduled visits

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
Change in loaded knee pain (single leg squat) visual analogue scale (VAS) | Baseline to 24 months post-surgery
  Used to demonstrate patient clinical improvement. The VAS is one of the most commonly used measures of pain intensity, where the patient rates their pain on a scale from 0 to 10 (0=no pain; 10=maximum pain possible).
Change in knee function measured by the TAS questionnaire | Baseline to 24 months post-surgery
  The TAS is a validated patient-administered questionnaire for use in multiple knee injuries and consists of a numerical scale ranging from 0 to 10 to indicate the ability to perform specific activities.
Change in knee function measured by the IKDC questionnaire | Baseline to 24 months post-surgery
  The IKDC measures the progress in symptoms, function, and sports activities caused by knee impairment after a treatment has been performed. It can be used with reliability and validity in patients with a range of knee conditions.
Change in knee function measured by the KOOS questionnaire | Baseline to 24 months post-surgery
  The KOOS is a measure of a patient's perceived knee pain and function, as well as associated problems with their knee status. It contains 42 items that are all recorded on a five-point Likert Scale by the patient.

SECONDARY OUTCOMES:
Repair tissue quantity and quality | Up to 24 months post-surgery
  Measured by MOCART Score and percentage lesion fill. The MOCART Score will be completed by two independent, blinded, well-trained radiologist readers.
Adverse events related to treatment | Up to 24 months post-surgery
Economic evaluation | surgical visit, 2 weeks, 6 weeks, 3 months, 6 months, 9 months,12 months and 24 months post-surgery
  Measured by study-specific Resource Utilization Questionnaires which will be used to determine the costs associated with the use of the BST-CarGel scaffold treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Desmarais, Study Chair — Piramal Healthcare Canada Ltd
Locations (15):
- Australia (2):
  - Calvary Wakefield Hospital, Adelaide
  - Murdoch Orthopaedic Clinic, Murdoch
- Canada (3):
  - Banff Sport Medicine, Banff
  - Fowler Kennedy Sport Medicine Clinic, London
  - Hôpital Maisonneuve-Rosemont, Montreal
- France (2):
  - Hopital de La Croix-Rousse, Lyon
  - CHRU Nancy - Hospital Central, Nancy
- University Medical Centre Regensburg, Regensburg, Germany
- Spain (4):
  - Hospital Universitari del Mar, Barcelona
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Miguel Servet, Zaragoza
- SportClinic Zurich / Hirslanden Clinic, Zurich, Switzerland
- United Kingdom (2):
  - The Royal Orthopaedic Hospital, Birmingham
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shive MS, Stanish WD, McCormack R, Forriol F, Mohtadi N, Pelet S, Desnoyers J, Methot S, Vehik K, Restrepo A. BST-CarGel(R) Treatment Maintains Cartilage Repair Superiority over Microfracture at 5 Years in a Multicenter Randomized Controlled Trial. Cartilage. 2015 Apr;6(2):62-72. doi: 10.1177/1947603514562064. PMID 26069709
- [Result] Stanish WD, McCormack R, Forriol F, Mohtadi N, Pelet S, Desnoyers J, Restrepo A, Shive MS. Novel scaffold-based BST-CarGel treatment results in superior cartilage repair compared with microfracture in a randomized controlled trial. J Bone Joint Surg Am. 2013 Sep 18;95(18):1640-50. doi: 10.2106/JBJS.L.01345. PMID 24048551